CLINICAL TRIAL: NCT01644448
Title: A Prospective Multicentric Open Label Randomized Bio-Interventional Phase I/II Pilot Study To Evaluate Safety & Efficacy Of Autologous Human Platelet Lysate (HPL) for Treatment of Periorbital Hyperpigmentation (Dark Circles)
Brief Title: A Study to Determine the Safety & Efficacy of Autologous Human Platelet Lysate (HPL) in Treatment of Dark Circles
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kasiak Research Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: KRPL/HPL-FR/11-12/002A
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Periorbital Hyperpigmentation (Dark Circles)
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study arm A (Other): Subjects will receive one dose of 5 ml of Autologous Human Platelet Lysate with simultaneous micro-needling on day 2
  Interventions: Other: Autologous Human Platelet Lysate
- Control Arm B (Other): Topical Applications of the standard therapy as directed by the investigator
  Interventions: Other: Standard Therapy

INTERVENTIONS:
Other: Autologous Human Platelet Lysate — Subjects will receive one dose of 5 ml of HPL with simultaneous micro-needling on day 2
  Arms: Study arm A
Other: Standard Therapy — Topical Applications as directed by the investigator
  Arms: Control Arm B

SUMMARY:
This is a multicentre, open label, randomized, pilot study to evalute safety and efficacy of Human Platelet Lysate (HPL) in subjects with Periorbital Hyperpigmentation. The study is being conducted at 2 centers in India.The primary endpoints are Physicians and Patient Self assessment score. The secondary endpoints are improvement in photographic assessment form randomization to end of study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (male and female), aged 18 to 55 years (both inclusive) with Periorbital Hyperpigmentation.
* Subject willing to refrain from any other treatment of Periorbital Hyperpigmentation during entire study duration.
* Subjects who are willing to give informed consent and adhere to the study protocol.

Exclusion Criteria:

* Subjects aged less than 18 and more than 55 years
* Subjects with history of connective tissue disease.
* Subjects with metabolic or hematopoietic disorders
* Subjects unwilling to or unable to comply with the study protocol.
* Subjects taking concomitant therapy that might interfere with the study results in the investigator's opinion or participating in another trial in the past 30 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-10 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Photographic Assessment | Day 0, Month 1, Month 2, End of Study - 3 months

OTHER OUTCOMES:
Physician's assessment scores | End of Study - 3 months
Patient's assessment scores | End of Study - 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Farida Modi, Dr., Principal Investigator — Dermacare; Preeti Savardekar, Dr., Principal Investigator — Shree Krishna Polyclinic; Sharmila Patil, Dr., Principal Investigator — Dr. Sharmila's Dermocosmetic laser center, hair and skin clinic
Locations (1):
- Kasiak Research Pvt Ltd, Thane, Maharashtra, India